CLINICAL TRIAL: NCT01838382
Title: Pain Characteristics After Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0871
Record Dates: First submitted 2013-04-16; First posted 2013-04-24 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Myoma of Uterus
Keywords: pain; total laparoscopic hysterectomy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- laparoscopic hysterectomy group (Experimental): female patients undergoing total laparoscopic hysterectomy.
  Interventions: Device: classic LMA insertion

INTERVENTIONS:
Device: classic LMA insertion — Classic LMA (cLMA) will be inserted when no response is obtained in the train-of-four stimulation. The fiberoptic view through the LMA, intraoperative complications of the cLMA, any complication during anesthesia emergence will be recorded. The device is examined and noted for the presence of visible blood.

SUMMARY:
Laparoscopic operative procedures have revolutionized gynecological surgery. These have several advantages: a smaller and more cosmetic incision, reduced blood loss and shorter postoperative stay, which cuts down on hospital costs. However, postoperative pain continues to be one complication, which results in an unpleasant experience for the patient and at times causes a delayed discharge. There are few studies about pain characteristics as one of laparoscopic hysterectomy complications. The purpose of this study is to investigate the prevalence and characteristics of shoulder pain, headache, abdominal pain, and back pain in patients undergoing total laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II
* age >=20, <= 80 years
* female
* patients undergoing elective total laparoscopic hysterectomy

Exclusion Criteria:

* age < 19 years or > 80 years
* abnormal mental status
* drug abuse
* chronic alcoholism
* immunosuppressants or steroid user

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
overall pain | 3 days
  evaluated with visual analogue score (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea